CLINICAL TRIAL: NCT01461291
Title: A Prospective, Randomized, Single-Masked, Controlled, Parallel Groups, Multicenter Clinical Investigation of the Glaukos® Trabecular Micro-Bypass Stent Model GTS400 Using the G2-M-IS Injector System in Conjunction With Cataract Surgery
Brief Title: Multicenter Study Using Glaukos® Trabecular Micro-Bypass Stent Model GTS400 Using the G2-M-IS Injector System in Conjunction With Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GC-008
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Primary open-angle glaucoma; POAG; Trabecular meshwork; iStent inject
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iStent inject (Experimental): Implantation of two GTS400 stents using G2-M-IS iStent inject
  Interventions: Device: iStent inject
- Cataract surgery (Active Comparator): Cataract surgery alone
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Device: iStent inject — Implantation of two GTS400 stents using G2-M-IS iStent inject
  Arms: iStent inject
Procedure: Cataract surgery — Cataract surgery alone
  Arms: Cataract surgery

SUMMARY:
Evaluate the safety and efficacy of the Glaukos Trabecular Micro-Bypass Stent Model GTS400 using the G2-M-IS injector system in conjunction with cataract surgery vs. cataract surgery only, in subjects with mild to moderate primary open-angle glaucoma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the Glaukos Trabecular Micro-Bypass Stent Model GTS400 using the G2-M-IS injector system in conjunction with cataract surgery, compared to cataract surgery only, in subjects with mild to moderate primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate open-angle glaucoma
* Characteristics consistent with mild/moderate glaucoma
* Use of one (1) to three (3) medications at time of screening exam

Exclusion Criteria:

* Pigmentary or pseudoexfoliative glaucoma
* Prior incisional glaucoma surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
≥ 20% Reduction in Intraocular Pressure (IOP) | Baseline and Month 24

SECONDARY OUTCOMES:
Diurnal IOP Reduction from Baseline | Baseline and Month 24

OTHER OUTCOMES:
Safety follow-up post-PMA to be through 36 months | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, O.D., Study Chair — Glaukos Corporation
Locations (1):
- Eye Centers of Racine and Kenosha, Racine, Wisconsin, United States